CLINICAL TRIAL: NCT05549388
Title: Effect of Front-of-Package Labels on the Intent to Purchase Packaged Foods in Ethiopia
Brief Title: Effect of Front-of-Pack Labels in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Addis Continental Institute of Public Health (Other); Resolve to Save Lives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00016498
Record Dates: First submitted 2022-09-02; First posted 2022-09-22 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Diseases
Keywords: Nutrition; Packaged food
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistical analyst will be masked to the study arms during the analysis phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No label (No Intervention): In this arm, participants will view images of packaged food or beverage products without a front-of-pack label and respond to questions about the products.
- Multiple Traffic Light (MTL) (Experimental): In this arm, participants will view images of packaged food or beverage products which have multiple traffic light labels displayed on the front-of-pack and respond to questions about the products.
  Interventions: Other: Front-of-pack labeling
- Nutri-Score (Experimental): In this arm, participants will view images of packaged food or beverage products which have a Nutriscore front-of-pack label and respond to questions about the products.
  Interventions: Other: Front-of-pack labeling
- Warning Label (Experimental): In this arm, participants will view packaged food or beverage products which have front-of-pack warning labels if the product is high in one or more nutrients of concern and respond to questions about the products.
  Interventions: Other: Front-of-pack labeling

INTERVENTIONS:
Other: Front-of-pack labeling — The intervention being tested is the effect of front-of-package labeling on consumers' intent to purchase foods which are high in one or more nutrients of public health concern. Participants randomized to the control group will view images of packaged foods and beverages and answer a series of questions about those products. In the intervention arms, participants will view images of the same packaged foods and beverages, but with different front-of-package labels displayed that provide nutrition information about the product. Participants in each arm will be asked the same series of questions about the products shown.
  Arms: Multiple Traffic Light (MTL); Nutri-Score; Warning Label

SUMMARY:
Ethiopia is experiencing the type of rapid food system transformation that leads to a double burden of malnutrition and increased non-communicable diseases. Front-of-pack labels on packaged foods are an emerging public health strategy with the potential to address non-communicable diseases by discouraging the purchase and consumption of products with high levels of nutrients of public health concern. The aim of this study is to evaluate and compare the effectiveness of front-of-pack labeling systems to reduce the intent to purchase unhealthy foods among adults in Ethiopia. The study will recruit approximately 1200 adults using a street-intercept methodology. Participants will be randomized to 1 of 4 arms to complete a survey in which the presence and type of front-of-pack label differs across survey arms and asked to rate participants' intent to purchase unhealthy packaged foods.

DETAILED DESCRIPTION:
In 2017, cardiovascular disease was the leading age-standardized cause of death in Ethiopia. The national prevalence of hypertension in Ethiopia in 2015 is estimated to be 16% (Gebreyes et al. 2018). Urban diets are rapidly changing, but not becoming healthier (Wolle et al. 2020). Diet quality remains poor: only 2.4% of the national population meets the WHO recommendation of five servings of fruit and vegetables per day. The mean estimated salt intake of 8.3 g/day exceeds the WHO maximum recommended intake (Challa et al. 2017). Processed foods are penetrating the market at a rapid pace (Melesse et al. 2019; Stuckler et al. 2012). Increasing income has increased demand for convenience foods (Minten et al. 2018). Ethiopia is experiencing the type of rapid food system transformation that leads to a double burden of malnutrition and increased non-communicable diseases (Popkin 2017).

Front-of-pack labels on packaged foods are an emerging public health strategy with the potential to address non-communicable diseases by discouraging the purchase and consumption of products with high levels of nutrients of public health concern (Croker et al. 2020). However, front-of-pack labels have not been tested in the Ethiopian context. Additionally, there are multiple types of front-of-pack labeling systems in use around the world, such as Multiple Traffic Light/Guideline Daily Amounts, the Nutri-Score system, and nutrient-specific warning labels.

Therefore, the study aims to to evaluate and compare the effectiveness of front-of-pack labeling systems to reduce the intent to purchase unhealthy foods among adults in Ethiopia. The study will recruit approximately 1200 adults using a street-intercept methodology. Participants will be randomized to 1 of 4 arms to complete a survey in which the presence and type of front-of-pack label differs across survey arms and asked to rate participants' intent to purchase unhealthy packaged foods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Purchase foods outside of the household

Exclusion Criteria:

* Age <18 years
* Do not purchase foods outside of the household
* Unable to complete the survey protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Intent to purchase based on single product tasks | The outcome will be assessed during survey administration at a single time point (baseline).
  Participants will be shown images of four single products, two of which are high in sodium and two of which are high in sugar. For each product, participants will rate their intent to purchase the product on a likert scale. The investigators will calculate the mean of the responses to questions about the four products.

SECONDARY OUTCOMES:
Purchase choice based on product comparison tasks | The outcome will be assessed during survey administration at a single time point (baseline).
  The investigators will evaluate responses to three product comparison tasks, each of which will present two packaged food items in the same food category and ask respondents which product they would choose to purchase. Specifically, the investigators will examine the proportion in each arm who report they would avoid purchasing the "less healthy" product.
Label understanding and acceptability | The outcome will be assessed during survey administration at a single time point (baseline).
  In the warning label, multiple traffic light, and Nutriscore arms, participants will be shown images of the respective labels. They will be asked a series of questions regarding their understanding of the label and its acceptability in Ethiopia and provide responses using a likert scale.

OTHER OUTCOMES:
Intent to purchase foods high in sodium | The outcome will be assessed during survey administration at a single time point (baseline).
  In exploratory analyses, the investigators will compare purchase intentions based on the single product tasks, examined separately for high sodium and high sugar products. For each product high in sodium, participants will rate their intent to purchase the product on a likert scale. The investigators will calculate the mean of the responses to questions about the two products high in sodium.
Intent to purchase foods high in sugar | The outcome will be assessed during survey administration at a single time point (baseline).
  In exploratory analyses, the investigators will compare purchase intentions based on the single product tasks, examined separately for high sodium and high sugar products. For each product high in sugar, participants will rate their intent to purchase the product on a likert scale. The investigators will calculate the mean of the responses to questions about the two products high in sugar.

CONTACTS AND LOCATIONS:
Locations (1):
- Street-Intercept Survey, Addis Ababa, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No
The investigators will only share deidentified data.

REFERENCES:
- [Background] Croker H, Packer J, Russell SJ, Stansfield C, Viner RM. Front of pack nutritional labelling schemes: a systematic review and meta-analysis of recent evidence relating to objectively measured consumption and purchasing. J Hum Nutr Diet. 2020 Aug;33(4):518-537. doi: 10.1111/jhn.12758. Epub 2020 May 4. PMID 32364292
- [Background] Popkin BM. Relationship between shifts in food system dynamics and acceleration of the global nutrition transition. Nutr Rev. 2017 Feb 1;75(2):73-82. doi: 10.1093/nutrit/nuw064. No abstract available. PMID 28395033
- [Background] Gebreyes YF, Goshu DY, Geletew TK, Argefa TG, Zemedu TG, Lemu KA, Waka FC, Mengesha AB, Degefu FS, Deghebo AD, Wubie HT, Negeri MG, Tesema TT, Tessema YG, Regassa MG, Eba GG, Beyene MG, Yesu KM, Zeleke GT, Mengistu YT, Belayneh AB. Prevalence of high bloodpressure, hyperglycemia, dyslipidemia, metabolic syndrome and their determinants in Ethiopia: Evidences from the National NCDs STEPS Survey, 2015. PLoS One. 2018 May 9;13(5):e0194819. doi: 10.1371/journal.pone.0194819. eCollection 2018. PMID 29742131
- [Background] Challa F, Tadesse Y, Mudie K, et al. Urinary Sodium Excretion and Determinants among Adults in Ethiopia: Findings from National STEPS Survey. Ethiopian Journal of Health Development. 2017; 31(1):370-77.
- [Background] Stuckler D, McKee M, Ebrahim S, Basu S. Manufacturing epidemics: the role of global producers in increased consumption of unhealthy commodities including processed foods, alcohol, and tobacco. PLoS Med. 2012;9(6):e1001235. doi: 10.1371/journal.pmed.1001235. Epub 2012 Jun 26. PMID 22745605
- See also: Melesse et al. 2019. Understanding urban consumers' food choice behavior in Ethiopia: Promoting demand for healthy foods. — http://www.ifpri.org/publication/understanding-urban-consumers%E2%80%99-food-choice-behavior-ethiopia-promoting-demand-healthy